CLINICAL TRIAL: NCT06407037
Title: Comparison of the Effects of Ultrasound-Guided Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block on Postoperative Acute Pain in Patients Undergoing Breast Surgery
Brief Title: Comparison of Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Arik, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2023-824
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Erector Spinae Plane Block; Serratus Posterior Superior Intercostal Plane Block; Acute Pain; Postoperative Pain; Breast Neoplasms
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 30 ml of 0.25% bupivacaine was injected into the area.
  Interventions: Procedure: Erector Spinae Plane Block
- Serratus Posterior Superior Intercostal Plane Block (Active Comparator): The probe was placed on the spinae scapula in the sagittal plane to identify the second and third ribs. The trapezius, rhomboid, serratus posterior superior muscle were visualized. The needle was inserted just above the third rib deeply into the serratus posterior superior muscle. Two mL isotonic was administrated for the correction. Then, 30 mL of 0.25% bupivacaine was administrated between serratus posterior superior muscle and rib.
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block will be performed unilaterally, under US guidance, before the surgical operation, when the patient is placed in the lateral decubitus position. 30 ml of 0.25% bupivacaine will be used in applications.
  Arms: Erector Spinae Plane Block
Procedure: Serratus Posterior Superior Intercostal Plane Block — Serratus Posterior Superior Intercostal Plane Block will be performed unilaterally, under US guidance, before the surgical operation, when the patient is placed in the lateral decubitus position. 30 ml of 0.25% bupivacaine will be used in applications.
  Arms: Serratus Posterior Superior Intercostal Plane Block

SUMMARY:
Breast cancer is the most common malignancy in women. Modified radical mastectomy, a surgical procedure in the treatment of breast cancer, is one of the standard treatments. Postoperative pain can seriously reduce the quality of life in patients, and inadequately treated acute pain can trigger chronic pain syndrome. Therefore, thoracic paravertebral block and thoracic epidural block are effective in postoperative analgesia. However, the use of these blocks is limited due to complications. In recent years, less invasive blocks, such as pectoral nerve block (PECS I-II), Serratus anterior plane block (SAPB), Erector spinae plane block (ESPB), and Serratus Posterior Superior intercostal Plane Block (SPSİPB) have been applied. In this study, it was aimed to compare the analgesic effectiveness of ESPB and SPSİPB applications in patients undergoing breast surgery.

DETAILED DESCRIPTION:
Postoperative pain will be assessed during resting and coughing with a visual analog scale (0-10 cm) and nausea and vomiting with a Postoperative Nausea Vomiting Score at the postoperative 1, 4, 8, 12, and 24 hours. The amount of tramadol consumed in the postoperative period will be recorded. Patient satisfaction will be assessed with the Likert scale at postoperative 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18-65
* Those with ASA scores I-II-III
* Those with a body mass index (BMI) between 18-35
* Patients who will undergo breast surgery

Exclusion Criteria:

* Those under the age of 18 and over the age of 65
* Those with ASA score IV and above
* Those with a history of allergy to the drugs to be blocked
* Those with a history of bleeding diathesis
* Patients with infection in the area to be blocked
* Those with a BMI below 18 and above 35
* Patients who underwent surgery under emergency conditions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | Postoperative day 1
  Pain will be assessed with a visual analog scale (0-10 cm)

SECONDARY OUTCOMES:
Postoperative tramadol consumption | Perioperative day 1
  The amount of tramadol consumed in the postoperative period will be recorded
Patient satisfaction | Postoperative 24th hour
  Satisfaction will be assessed with a 5 point Likert scale (0-4 whereas 0:definitely disagree; 1:slightly agree; 3: agree; 4: strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)